CLINICAL TRIAL: NCT02769104
Title: Aromatase Inhibitors (AI) Plus Chemotherapy Versus Chemotherapy as Neoadjuvant Treatment in Postmenopausal Hormone Receptor-positive Breast Cancer
Brief Title: Aromatase Inhibitors Plus Chemotherapy vs Chemotherapy as Neoadjuvant Treatment in Postmenopausal HR(+) Breast Cancer
Acronym: ACCN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZJCH-ACCN
Record Dates: First submitted 2016-05-08; First posted 2016-05-11 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Neoadjuvant Therapy
Keywords: aromatase inhibitors; chemotherapy; neoadjuvant; postmenopausal; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Aromatase Inhibitors; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AI+Chemo (Experimental): aromatase inhibitors (Letrozole 2.5mg po. QD for 5 years) starts at the beginning of neoadjuvant treatment combined with chemotherapy (AC*4-T*4) in patients with postmenopausal hormone receptor-positive breast cancer
  Interventions: Drug: Letrozole (Aromatase Inhibitors); Drug: AC*4-T*4
- Chemo (Active Comparator): chemotherapy (AC*4-T*4) as neoadjuvant treatment without aromatase inhibitors in patients with postmenopausal hormone receptor-positive breast cancer
  Interventions: Drug: AC*4-T*4

INTERVENTIONS:
Drug: Letrozole (Aromatase Inhibitors) — Letrozole (Aromatase Inhibitors) for 5 years
  Other Names: Letrozole
  Arms: AI+Chemo
Drug: AC*4-T*4 — CTX800mg/m2 d1+Anthracyclines75mg/m2 d1, every 3 weeks*4 cycles, be sequential with Docetaxel 75mg/m2 d1, every 3 weeks*4cycles
  Other Names: CTX+Anthracyclines, Docetaxel

SUMMARY:
The investigators designed this study to investigate the effect of aromatase inhibitors (AI) plus chemotherapy versus chemotherapy as neoadjuvant treatment in postmenopausal hormone receptor-positive breast cancer.

DETAILED DESCRIPTION:
The endocrine therapy has been used more and more in neoadjuvant treatment of hormone receptor-positive breast cancer. But it still a question if neoadjuvant endocrine therapy can be used combined with chemotherapy. There have been several small-sample studies concerning about this item and also got some results that support the suppose that endocrine therapy combined with chemotherapy could rise the effect of neoadjuvant treatment. This study is to investigate the effect of aromatase inhibitors (AI) plus chemotherapy versus chemotherapy as neoadjuvant treatment in postmenopausal hormone receptor-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* provision of informed consent
* clinical stage IIA~IIIC
* histologically proven HR+ invasive breast cancer
* women defined as postmenopausal according to NCCN guideline
* plan to accept the neoadjuvant (pre operational) chemotherapy treatment

Exclusion Criteria:

* clinical evidence of metastatic disease
* bilateral oophorectomy;
* radiation of the ovaries
* patients who, for whatever reason (e.g., confusion, infirmity, alcoholism), are unlikely to comply with trial requirements
* patients who accepted anti-cancer treatment before
* previous hormonal therapy as adjuvant treatment for non-cancer disease
* patients unwilling to stop taking any drug known to affect sex hormonal status, or in whom it would be inappropriate to stop
* previous history of invasive malignancy within the last 5 years, other than squamous or basal cell carcinoma of the skin or carcinoma in situ of the cervix, adequately cone biopsied
* treatment with a non-approved or experimental drug during 1 month before entry into the study
* history of bleeding diathesis (i.e., Disseminated intravascular coagulation, clotting factor deficiency), or long term anticoagulant therapy (other than antiplatelet therapy and low dose warfarin)
* leukopenia and/or thrombocytopenia
* history of ocular fundus diseases
* history of thromboembolic diseases
* history of osteoporotic fractures

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
effective rate | half year after randomized
  CR+PR

SECONDARY OUTCOMES:
pCR | half year after randomized
  pathological CR
disease-free survival (DFS) | 2 years after randomized
  disease-free survival
side effect rate | 2 years after randomized

CONTACTS AND LOCATIONS:
Overall Officials: Hong-Jian Yang, MD., Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
The investigators have not decided if the data can be available.